CLINICAL TRIAL: NCT00310960
Title: An Observational Study of Infantile, Acquired Non-accommodative, and Acquired Partially-accommodative Esotropia
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NEI-102; 2U10EY011751 (NIH); 5U10EY011751 (NIH)
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Infantile Esotropia; Acquired Non-accommodative Esotropia; Acquired Partially Accommodative Esotropia
Keywords: infantile esotropia; acquired non-accommodative esotropia; acquired partially accommodative esotropia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to:

* To estimate the duration of misalignment by age at presentation in infantile esotropia (infantile ET), acquired non-accommodative esotropia (ANAET) and acquired partially accommodative esotropia (APAET).
* To determine the proportion of patients with angle instability in infantile ET, ANAET and APAET by length of follow-up.

DETAILED DESCRIPTION:
Approximately one third of infants with infantile esotropia (infantile ET) and a similar proportion of children with acquired non-accommodative esotropia (ANAET) will have an increasing angle within the first few months of their initial examination. In approximately two thirds of patients, the angle of misalignment remains stable and in a small proportion, the angle of esotropia decreases. The changing angle of misalignment in a significant proportion of children with esotropia raises an important question regarding the timing of surgical management of these children: should surgery be undertaken immediately or delayed until the alignment stabilizes? Early surgery may improve sensory outcomes; delayed surgery may improve surgical dosing accuracy and motor outcomes.

Children with acquired partially accommodative esotropia (APAET) may differ from those with infantile ET and ANAET in that they tend to present at an older age, are more likely to preserve high-grade stereopsis with appropriate treatment, require surgical intervention less frequently, and have more substantial hyperopic refractive errors. Little is known regarding early angle stability in this group of patients following correction of their refractive errors.

Although there is a need for a randomized trial to address the issue of timing of surgery in infantile ET, APAET, and ANAET, prior to designing such a trial, high-quality preliminary data are needed. We propose a multi-center observational study to 1) determine the duration of misalignment in infantile ET, ANAET, and APAET at study enrollment, 2) to prospectively establish the proportion of patients with angle instability in infantile ET, ANAET, and APAET, and 3) to determine recruitment potential for a randomized trial. These data will be crucial for sample size calculations for the eventual randomized trial, and will help further define the clinical characteristics of these conditions.

A concurrent and nested ancillary study will be conducted at selected centers to collect test-retest data on alignment measurements for estimating the amount of measurement variability. These test-retest data will be used to define a change in angle alignment that exceeds an amount which could reasonably be due to measurement error, which will be used in evaluating the proportion of patients with angle instability in the current study.

Eligible patients with infantile ET will be consented and enrolled at their initial visit. Infantile ET patients who need spectacles will be prescribed spectacles and will return for an Infantile ET Spectacle Baseline Visit 2 weeks later.

ANAET and APAET patients who present wearing spectacles with appropriate correction for at least 2 weeks will be consented and enrolled into the study at that initial visit.

For ANAET and APAET patients who present not wearing spectacles:

* Patients who do not need spectacles will be consented and enrolled into the study at that initial visit.
* Patients who need spectacles are prescribed appropriate correction if the investigator intends to offer the patient enrollment at a later date. Patients are asked to return after wearing the new spectacles 2-6 weeks, at which time they may be consented and enrolled into the study.

Sample Size: The study will enroll 100 patients for each of the three esotropia types of infantile ET, ANAET, and APAET, for a total of 300 patients.

ELIGIBILITY:
Inclusion Criteria:

For infantile ET:

* Less than 12 months old
* Duration of esotropia less than 6 months by best estimate (photos, parent history, physician records)
* A constant or variable esotropia
* Onset before six months of age
* Measuring >10 PD by Alternate Prism and Cover Test (APCT) in the primary position at distance fixation on an accommodative target
* Gestational age > 34 weeks
* Birth weight > 1500 grams

For ANAET:

* 6 months to <5 years old
* Duration of esotropia less than 6 months by best estimate (photos, parent history, physician records)
* A constant or variable esotropia
* Onset after six months of age
* Angle decreases less than 10 prism diopters (PD) by Alternate Prism and Cover Test (APCT) in the primary position at distance fixation with correction
* Residual angle measures >10 PD by Simultaneous Prism and Cover Test (SPCT) in the primary position at distance fixation
* For patients who have significant refractive error, full hyperopic correction determined with cycloplegia must have been worn for at least 2 weeks.
* For patients who do not have significant refractive error, whether to prescribe spectacles is at investigator discretion, however, if the investigator elects to prescribe spectacles, the full hyperopic correction determined with cycloplegia must have been worn for at least 2 weeks
* Gestational age > 34 weeks
* Birth weight > 1500 grams

For APAET:

* Onset after six months of age
* 6 months to <5 years old
* Duration of esotropia less than 6 months by best estimate (photos, parent history, physician records)
* Angle decreases 10 prism diopters (PD) or more by Alternate Prism and Cover Test (APCT) in the primary position at distance fixation with correction
* A constant or variable esotropia
* Residual angle measures >10 PD by Simultaneous Prism and Cover Test (SPCT) in the primary position at distance fixation
* For patients who have significant refractive error, full hyperopic correction determined with cycloplegia must have been worn for at least 2 weeks.
* For patients who do not have significant refractive error, whether to prescribe spectacles is at investigator discretion, however, if the investigator elects to prescribe spectacles, the full hyperopic correction determined with cycloplegia must have been worn for at least 2 weeks
* Gestational age > 34 weeks
* Birth weight > 1500 grams

Exclusion Criteria:

For infantile ET:

* prior spectacle wear

For infantile ET,ANAET,APAET:

* Atropine use within the last two weeks
* History of CNS disease (e.g. intraventricular hemorrhage (IVH), PVL, meningitis, developmental abnormalities of the brain, hydrocephalus, cerebral palsy, hypoxic ischemic encephalopathy)
* Significant developmental delay in the investigator's judgment (isolated speech delay excepted)
* Limitation of abduction consistent with paralytic or restrictive myopathy (minor limitation of abduction due to cross fixation is acceptable)
* Craniofacial malformation affecting the orbits
* Prior extraocular muscle surgery or intraocular surgery
* Structural ocular abnormalities (e.g. media opacity, optic atrophy, optic nerve hypoplasia, retinal detachment)

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2004-06; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Determination of angle instability | 18 weeks
Estimation of misalignment | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P. Christiansen, M.D., Study Chair — University of Minnesota
Locations (1):
- University of Minnesota Medical School, Minneapolis, Minnesota, United States